CLINICAL TRIAL: NCT06743685
Title: A Pilot Feasibility Trial of HEALthy Beginnings: A Trauma-Informed, Chronic Disease Self-Care Intervention for Middle-Aged, and Older Homeless Women
Brief Title: Pilot Feasibility Trial of HEALthy Beginnings for Middle-Aged, and Older Homeless Women
Acronym: HB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Hillman Foundation (Unknown)
Responsible Party: Principal Investigator, Benissa E. Salem, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-001117; 85834 (Other Grant/Funding Number: Hillman)
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Homelessness; Health Promotion; Chronic Disease Self-care; Multimorbidity; Unhoused
Keywords: Middle-aged and older; People experiencing homelessness; Women; Elderly; Trauma-informed care

STUDY DESIGN:
Intervention Model Description: All eligible participants will be invited to enroll in the HEALthy Beginnings intervention, a trauma-informed, chronic disease self-care intervention for middle-aged, and older homeless women. Participants will attend nine group sessions and six individual sessions over approximately 12 weeks. A subset of participants will be invited to participate in post-intervention focus groups as well as to complete a questionnaire evaluating the HEALthy Beginnings intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HEALthy Beginnings Intervention group (Experimental): Middle-aged, and older, homeless women (MAO-HW) participating in the HEALthy Beginnings Intervention
  Interventions: Behavioral: HEALthy Beginnings

INTERVENTIONS:
Behavioral: HEALthy Beginnings — HEALthy Beginnings, an innovative, enhanced, trauma-informed, chronic disease self-care program and nurse-driven intervention, developed and tailored for middle-aged, and older, homeless women (MAO-HW).

SUMMARY:
This is a mixed methods pilot feasibility trial of HEALthy Beginnings, an innovative, nurse-driven intervention. Middle-aged and older, homeless women (MAO-HW) will participate in the HEALthy Beginnings intervention and select MAO-HW will be invited to participate in post-intervention qualitative focus groups to evaluate the program.

DETAILED DESCRIPTION:
This pilot feasibility trial will enroll middle-aged and older, homeless women (MAO-HW) in the HEALthy Beginnings intervention. Participants will be asked to complete a baseline questionnaire and locator guide. Participants will then engage over a period of approximately three months in nine 60-90 minute group sessions focused on health topics, and to meet with a research team member for six private sessions which will last up to 45 minutes each to assess the program and discuss content.

Fifteen participants will be asked to return at completion of the group/individual sessions to participate in a post-intervention qualitative focus group and follow-up questionnaire to evaluate the HEALthy Beginnings intervention.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported age 40 years or older
* Sex assigned Female at birth
* Homeless, or living in a shelter designed to provide transitional housing
* Self-reported multimorbidity (at least 2 physical/mental health conditions)
* Able to communicate in English

Exclusion Criteria:

* Experiencing hallucinations
* Exhibiting signs of acute intoxication (e.g., slurred speech, pin-point pupils, difficulty walking)
* Non-English speaking
* Unable to understand study procedures (e.g., screening questions)

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Recruitment as a measure of feasibility of the HEALthy Beginnings intervention | Day 1
  Number of eligible participants who enroll in the program after screening
Completion as a measure of feasibility of the HEALthy Beginnings intervention | Upon completion of all group and individual sessions, approximately 12 Weeks
  Number of enrolled participants who complete the intervention

SECONDARY OUTCOMES:
Participant evaluation of HEALthy beginnings intervention | Upon completion of all group and individual sessions, approximately 12 Weeks
  HEALthy Beginnings will be evaluated by post-intervention focus group participants via a questionnaire consisting of 12 questions in 3 subscales. Response to each question is a 5-point Likert scale, with a score range of 12-60 points for an overall representation of acceptability, appropriateness & feasibility. Higher scores indicate more favorable evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Benissa E. Salem, PhD, MSN, RN, CNL, PHN, Principal Investigator — University of California, Los Angeles
Locations (1):
- Downtown Women's Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No